CLINICAL TRIAL: NCT03333915
Title: An Open Label, Multi-Center Phase I/II Study to Evaluate Efficacy and Safety of BGB-290 in Chinese Subjects With Advanced Ovarian Cancer, Fallopian Cancer, and Primary Peritoneal Cancer or Advanced Triple Negative Breast Cancer
Brief Title: Study of the Efficacy, Safety and Pharmacokinetics of Pamiparib (BGB-290) in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-290-102; CTR20160828 (Registry Identifier: ChiCTR)
Record Dates: First submitted 2017-11-01; First posted 2017-11-07 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2023-07

CONDITIONS: Advanced High-grade Ovarian Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pamiparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1: 20 milligram (mg) pamiparib (Experimental): 20 mg pamiparib twice a day for 21 days
  Interventions: Drug: Pamiparib
- Phase 1 : 40 mg pamiparib (Experimental): 40 mg pamiparib twice a day for 21 days
  Interventions: Drug: Pamiparib
- 60 mg pamiparib (Experimental): 60 mg pamiparib twice a day for 21 days
  Interventions: Drug: Pamiparib
- 60 mg pamiparib in platinum-sensitive ovarian cancer (PSOC) (Experimental): 60 mg pamiparib twice a day until occurrence of unacceptable toxicities, disease progression, withdrawal of consent or investigator discretion
  Interventions: Drug: Pamiparib
- 60 mg pamiparib in platinum resistant ovarian cancer (PROC) (Experimental): 60 mg pamiparib twice a day until occurrence of unacceptable toxicities, disease progression, withdrawal of consent or investigator discretion
  Interventions: Drug: Pamiparib

INTERVENTIONS:
Drug: Pamiparib — Pamiparib is provided as oral capsules
  Other Names: BGB-290

SUMMARY:
This study is designed to evaluate the safety, tolerability, PKharmacokinetic profile and treatment effect of pamiparib in Chinese participants with advanced high-grade ovarian cancer (including fallopian cancer or primary peritoneal cancer) and triple negative breast cancer in phase I, and to evaluate the efficacy and safety of pamiparib in Chinese participants with recurrent epithelial ovarian cancer (including fallopian cancer or primary peritoneal cancer), harboring germline breast cancer susceptibility gene 1/gene 2 (BRCA1/2) mutation in phase II.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants have voluntarily agreed to participate by giving written informed consent.
2. Age 18 years (including 18 years) on the day of signing informed consent.
3. Participants meet the following eligibility criteria for the corresponding part of the study: 1) In Phase 1 portion: The participants must have a histologically or cytologically confirmed locally advanced or metastatic cancer, either triple-negative breast cancer or epithelial, non-mucinous, high-grade ovarian cancer (including fallopian cancer, or primary peritoneal cancer), for which no effective standard therapy is available.

2) In Phase 2 portion: Participants who have histologically or cytologically confirmed high-grade epithelial ovarian cancer (including fallopian cancer or primary peritoneal cancer), harboring germline BRCA1/2 mutation 4. Participants must have measurable disease as defined per the RECIST, version 1.1.

5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1

Key Exclusion Criteria:

1. Participants who have been treated with chemotherapy, biologic therapy, immunotherapy, investigational agent, anti-cancer Chinese medicine, or anticancer herbal remedies ≤ 14 days (or ≤5 half-lives, whichever is shorter) prior to starting study drug, or who have not adequately recovered from the side effects of such therapy.
2. Participants who have undergone major surgery for any cause ≤ 4 weeks prior to starting study drug. Participants must have adequately recovered from the previous treatment and have a stable clinical condition before entering the study.
3. Participants who have undergone radiotherapy for any cause ≤ 14 days prior to starting study drug. Participants must have adequately recovered from the previous treatment and have a stable clinical condition before entering the study.
4. Untreated and/or active brain metastases.
5. Prior therapies targeting poly (ADP-ribose) polymerase (PARP).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (6):
- China (6):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 2 Phases. Phase 1 (December 2016 to December 2019) in which 15 participants were enrolled and Phase 2 (December 2017 to August 2021) in which 113 participants were enrolled. Primary data cut off date for Phase 1 was 24 December 2019 and Primary cut-off date for Phase 2 was 24 August 2020.
Groups:
- Phase 1: 20 Milligram (mg) Pamiparib: Participants received a single dose of 20 mg pamiparib orally on Day 1 followed by one day treatment free period (Day 2), and 20 mg pamiparib twice a day for the following 21 days (Day 3 to Day 23) until unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
- Phase 1: 40 mg Pamiparib: Participants received a single dose of 40 mg pamiparib orally on Day 1 followed by one day treatment free period (Day 2), and 40 mg pamiparib twice a day for the following 21 days (Day 3 to Day 23) until unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
- Phase 1: 60 mg Pamiparib: Participants received a single dose of 60 mg pamiparib orally on Day 1 followed by a one day treatment free period (Day 2), and 60 mg pamiparib twice a day for the following 21 days (Day 3 to Day 23) until unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
- Phase 2: 60 mg Pamiparib in Platinum-sensitive Ovarian Cancer (PSOC): Participants with PSOC received 60 mg pamiparib twice a day on Day 1 of Cycle 1 (21-day cycle) and continuously in all subsequent cycles until occurrence of unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
- Phase 2: 60 mg Pamiparib in Platinum-resistant Ovarian Cancer (PROC): Participants with PROC received 60 mg pamiparib twice a day on Day 1 of Cycle 1 (21-day cycle) and continuously in all subsequent cycles until occurrence of unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
Period: Overall Study
Arm/Group | Phase 1: 20 Milligram (mg) Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib | Phase 2: 60 mg Pamiparib in Platinum-sensitive Ovarian Cancer (PSOC) | Phase 2: 60 mg Pamiparib in Platinum-resistant Ovarian Cancer (PROC)
Started | 4 | 4 | 7 | 90 | 23
Completed | 4 | 3 | 6 | 0 | 0
Not Completed | 0 | 1 | 1 | 90 | 23
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 37 | 18
Not completed — Sponsor's Decision | 0 | 0 | 0 | 48 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set includes all participants who received at least one dose of pamiparib
Groups:
- Phase 1: 20 mg Pamiparib: Participants received a single dose of 20 mg pamiparib orally on Day 1 followed by one day treatment free period (Day 2), and 20 mg pamiparib twice a day for the following 21 days (Day 3 to Day 23) until unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
- Phase 2: 60 mg Pamiparib in PSOC: Participants with PSOC received 60 mg pamiparib twice a day on Day 1 of Cycle 1 (21-day cycle) and continuously in all subsequent cycles until occurrence of unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
- Phase 2: 60 mg Pamiparib in PROC: Participants with PROC received 60 mg pamiparib twice a day on Day 1 of Cycle 1 (21-day cycle) and continuously in all subsequent cycles until occurrence of unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
- Total: Total of all reporting groups
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC | Total
Number analyzed (Participants) | 4 | 4 | 7 | 90 | 23 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (6.55) | 48.0 (13.95) | 53.0 (9.15) | 54.4 (7.94) | 52.9 (7.97) | 53.87 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 7 | 90 | 23 | 128
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 7 | 90 | 23 | 128
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 4 | 7 | 90 | 23 | 128

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Treatment- Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE)
Description: A TEAE is defined as an adverse event (AE) that had an onset date on or after the first dose of study drug up to 30 days following study drug discontinuation or was worsening in severity from baseline (pretreatment).
Time Frame: From first dose to within 30 days of last dose of pamiparib (approximately 36 months)
Population: Safety Analysis Set includes all participants who received at least one dose of pamiparib
Measure: Number; unit: Number of participants
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 7
Number of participants
  Participants with at least 1 TEAE | 4 | 4 | 7
  Treatment-Emergent SAEs | 0 | 1 | 2

2. Primary Outcome: Phase 1: Number of Participants With Clinically Significant Abnormalities in Physical Examinations and Electrocardiograms (ECGs)
Time Frame: From first dose to within 30 days of last dose of pamiparib (approximately 36 months)
Population: Safety Analysis Set
Measure: Number; unit: Number of participants
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 7
Number of participants
  Physical Findings | 0 | 0 | 0
  ECGs | 0 | 0 | 0

3. Primary Outcome: Phase 2: Objective Response Rate (ORR) in High Grade Ovarian Cancer (HGOC) Both PSOC and PROC as Assessed by Independent Radiology Review Committee (IRC)
Description: ORR is defined as the percentage of participants with confirmed Complete Response or Partial Response
Time Frame: Up to approximately 2 years and 8 months
Population: Efficacy Evaluable Set defined as all participants in the Safety Analysis Set who had measurable disease at baseline per RECIST v1.1. participants with available data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC
Number analyzed (Participants) | 82 | 19
Percentage of participants | 68.3 [57.1 to 78.1] | 31.6 [12.6 to 56.6]

4. Secondary Outcome: Phase I: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Cycle 1 Day 1 and Day 10 of 21-day cycle: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: PK Analysis Set was defined as all participants for whom valid PK parameters could be estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 7
ng/mL
  Day 1 | 718.4 (18.9) | 1633.7 (12.2) | 2302.5 (30.1)
  Day 10 | 1280.1 (70.5) | 5213.8 (25.6) | 5861.3 (29.2)

5. Secondary Outcome: Phase I: Time to Reach Cmax (Tmax)
Time Frame: Cycle 1 Day 1 and Day 10 of 21-day cycle: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: PK Analysis Set
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 7
hours
  Day 1 | 1.01 [0.52 to 3.78] | 0.98 [0.97 to 1.05] | 1.13 [1.00 to 6.08]
  Day 10 | 1.04 [0.92 to 2.12] | 1.10 [0.98 to 1.95] | 1.13 [0.98 to 1.97]

6. Secondary Outcome: Phase I: Terminal Elimination Half-life (t1/2)
Time Frame: Cycle 1 Day 1 of 21-day cycle: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: PK Analysis Set
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 7
hours | 12.14 [8.15 to 18.15] | 11.79 [8.74 to 20.14] | 13.77 [6.54 to 34.91]

7. Secondary Outcome: Phase I: Apparent Clearance (CL/F)
Time Frame: Cycle 1 Day 1 of 21-day cycle: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 7
Liters/hour (L/h) | 1.95 (43.85) | 2.07 (61.09) | 2.19 (79.41)

8. Secondary Outcome: Phase 1: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUCinf)
Time Frame: Cycle 1 Day 1 of 21-day cycle: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: Pharmacokinetic (PK) Analysis Set includes all participants for whom valid pamiparib PK parameters could be estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter (h*ng/mL)
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 7
Hours*nanograms/milliliter (h*ng/mL) | 1020.5 (43.9) | 1912.7 (61.1) | 27454.4 (79.4)

9. Secondary Outcome: Phase I: Apparent Volume of Distribution During Terminal Phase (Vz/F)
Time Frame: Cycle 1 Day 1 of 21-day cycle: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 7
Liters | 34.2 (23.6) | 35.2 (21.8) | 37.2 (33.2)

10. Secondary Outcome: Phase I: Confirmed Objective Response Rate (ORR) as Assessed by the Investigator Per RECIST v1.1
Description: ORR is defined as the percentage of participants with confirmed Complete Response (CR) or Partial Response (PR)
Time Frame: Up to approximately 36 months
Population: Efficacy Evaluable Set includes all participants in the safety analysis set who had the measurable disease at baseline per RECIST v1.1 and had at least one post-baseline tumor assessment unless discontinued due to clinical progression or death prior to assessment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 5
Percentage of participants | 25.0 [0.6 to 80.6] | 25.0 [0.6 to 80.6] | 0 [0.0 to 52.2]

11. Secondary Outcome: Phase 1: Disease Control Rate (DCR) Assessed by the Investigator Per RECIST v1.1
Description: DCR is defined as the percentage of participants with best overall response (BOR) of CR, PR and stable disease (SD)
Time Frame: Up to approximately 36 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 5
Percentage of participants | 50.0 [6.3 to 93.2] | 50.0 [6.8 to 93.2] | 80.0 [28.4 to 99.5]

12. Secondary Outcome: Phase I: Clinical Benefit Rate (CBR) Assessed by the Investigator Per RECIST v1.1
Description: CBR is defined as percentage of participants with best overall response of CR, PR and stable disease (SD)≥24 weeks
Time Frame: Up to approximately 36 months
Population: Efficacy Evaluable Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 5
Percentage of participants | 25.0 [0.6 to 80.6] | 50.0 [6.8 to 93.2] | 40.0 [5.3 to 85.3]

13. Secondary Outcome: Phase 1: Duration of Response (DOR) as Assessed by Investigator Per RECIST v1.1
Description: DOR is defined as the time from the first determination of a confirmed overall response until the first documentation of progression or death, whichever comes first
Time Frame: Up to approximately 36 months
Population: Efficacy Evaluable Set; Only the number of responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 1 | 1 | 0
months | 30.4 [NA to NA] — NA = Not estimable due to insufficient number of events | NA [NA to NA] — NA = Not estimable due to insufficient number of events |

14. Secondary Outcome: Phase I : Progression Free Survival (PFS)
Description: PFS is defined as the time from first dose of study medication to the first documented disease progression or death due to any cause, whichever occurs first
Time Frame: Up to approximately 36 months
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib
Number analyzed (Participants) | 4 | 4 | 7
Months | 2.2 [1.48 to 34.53] | NA [1.45 to NA] — NA = Not estimable due to insufficient number of events | 5.6 [1.48 to NA] — NA = Not estimable due to insufficient number of events

15. Secondary Outcome: Phase 2: Objective Response Rate (ORR) by Investigator Per RECIST v1.1
Description: ORR is defined as the percentage of participants with confirmed Complete Response or Partial Response
Time Frame: Up to approximately 3 years and 8 months
Population: Efficacy Analysis Set; Participants with available data were included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC
Number analyzed (Participants) | 82 | 19
Percentage of participants | 64.6 [53.3 to 74.9] | 26.3 [9.1 to 51.2]

16. Secondary Outcome: Phase 2: Disease Control Rate by Investigator Per RECIST v1.1
Description: DCR is defined as the percentage of participants with best overall response (BOR) of CR, PR and stable disease (SD)
Time Frame: Up to approximately 3 years and 8 months
Population: Efficacy Analysis Set; Participants with available data were included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC
Number analyzed (Participants) | 90 | 23
Percentage of participants | 96.3 [89.7 to 99.2] | 78.9 [54.4 to 93.9]

17. Secondary Outcome: Phase 2: Clinical Benefit Rate by Investigator Per RECIST v1.1
Description: CBR is defined as percentage of participants with best overall response of CR, PR and stable disease (SD)≥24 weeks
Time Frame: Up to approximately 3 years and 8 months
Population: Efficacy Analysis Set; Participants with available data were included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC
Number analyzed (Participants) | 90 | 23
Percentage of participants | 73.2 [62.2 to 82.4] | 52.6 [28.0 to 75.6]

18. Secondary Outcome: Phase 2: Carcinoma Antigen-125 (C(A-125) Response Rate by Gynecologic Cancer Inter Group (GCIG )Criteria
Description: CA-125 response is defined the percentage of participants with at least 50% reduction in CA-125 levels from pre-treatment sample
Time Frame: Up to approximately 3 years and 8 months
Population: CA-125 Evaluable Analysis Set is defined as a subset of participants in the Safety Analysis with baseline CA-125 >/= 2 X upper limit of normal (ULN)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC
Number analyzed (Participants) | 90 | 23
Percentage of participants | 79.7 [68.8 to 88.2] | 38.1 [18.1 to 61.8]

19. Secondary Outcome: Phase 2: Duration of Response as Assessed by Investigator Per RECIST v1.1
Description: as for outcome 13
Time Frame: Up to approximately 3 years and 8 months
Population: Efficacy Evaluable Set : Participants with available data were included in the analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC
Number analyzed (Participants) | 82 | 19
Months | 11.1 [9.00 to 14.52] | 6.9 [4.93 to 19.78]

20. Secondary Outcome: Phase 2: Progression Free Survival as Assessed by the Investigator Per RECIST v1.1
Description: as for outcome 14
Time Frame: Up to approximately 3 years and 8 months
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC
Number analyzed (Participants) | 90 | 23
Months | 10.4 [8.31 to 15.15] | 5.5 [2.27 to 6.24]

21. Secondary Outcome: Phase 2: Overall Survival (OS) as Assessed by Investigator
Description: OS is defined as time from the first dose of study medication to the date of death due to any cause
Time Frame: Up to approximately 3 years and 8 months
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC
Number analyzed (Participants) | 90 | 23
Months | 34.1 [29.08 to NA] — NA = Not estimable due to insufficient number of events | 13.6 [7.13 to 19.75]

22. Secondary Outcome: Phase 2: Number of Participants With Treatment- Emergent Adverse Events and Serious Adverse Events
Description: A TEAE is defined as an adverse event (AE) that had an onset date on or after the first dose of study drug up to 30 days following study drug discontinuation or was worsening in severity from baseline (pretreatment). All clinically significant abnormalities in physical examinations, laboratory tests and ECGs are reported as adverse events (AE) in the AE section.
Time Frame: From first dose to within 30 days of last dose of pamiparib (approximately 3 years and 8 months)
Population: Safety Analysis Set
Measure: Number; unit: Number of participants
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC | Phase 2: 60 mg Pamiparib in PROC
Number analyzed (Participants) | 90 | 23
Number of participants
  Participants With At Least one TEAE | 90 | 23
  Treatment Emergent SAEs | 36 | 15

23. Secondary Outcome: Phase 2: Area Under the Plasma Concentration-time Curve From 0 to 12 Hours Post-dose (AUC0-12)
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: PK Analysis Set: Participants with at least one available PK parameter at the specified visit were included in the analysis. Phase 2 PK analyses were performed for all Phase 2 participants combined per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter (h*ng/mL)
Groups:
- Phase 2: 60 mg Pamiparib in PSOC or PROC: Participants with PSOC or PROC received 60 mg pamiparib twice a day on Day 1 of Cycle 1 (21-day cycle) and continuously in all subsequent cycles until occurrence of unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC or PROC
Number analyzed (Participants) | 15
hours*nanograms/milliliter (h*ng/mL)
  Cycle 1 Day 1 | 16841.5 (20.5)
  Cycle 2 Day 1: number analyzed (Participants) | 12
  Cycle 2 Day 1 | 48802.4 (24.3)

24. Secondary Outcome: Phase 2: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC or PROC
Number analyzed (Participants) | 15
ng/mL
  Cycle 1Day 1 | 2275.1 (19.6)
  Cycle 2 Day 1: number analyzed (Participants) | 12
  Cycle 2 Day 1 | 5251.5 (22.7)

25. Secondary Outcome: Phase 2: Time to Reach Cmax (Tmax)
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: as for outcome 23
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC or PROC
Number analyzed (Participants) | 15
hours
  Cycle 1 Day 1 | 1.88 [0.95 to 3.98]
  Cycle 2 Day 1: number analyzed (Participants) | 12
  Cycle 2 Day 1 | 1.98 [0.50 to 4.00]

26. Secondary Outcome: Phase 2: Area Under the Plasma Concentration-time Curve From 0 to the 9 Hours Post-dose (AUC0-9)
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1: pre-dose, 0.5, 1, 2, 4, 6,9 and 12 hours post dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 2: 60 mg Pamiparib in PSOC or PROC
Number analyzed (Participants) | 15
h*ng/mL
  Cycle 1 Day 1 | 13577.2 (20.3)
  Cycle 2 Day 1: number analyzed (Participants) | 12
  Cycle 2 Day 1 | 38259.3 (23.5)

ADVERSE EVENTS:
Time Frame: Phase1: From first dose to within 30 days of last dose of pamiparib (approximately 36 months) Phase 2: From first dose to within 30 days of last dose of pamiparib (approximately 3 years and 8 months)
Description: Adverse Events were coded based on MedDRA version 22.0 for Phase 1, and version 24.0 for Phase 2. All clinically significant abnormalities in physical examinations, laboratory tests and ECGs in Phase 1 and Phase 2 are reported as adverse events.
Groups:
- Phase 1: 20 mg Pamiparib: Participants received a single dose of 20 mg pamiparib orally on Day 1 followed by a one day treatment free period (Day 2), and 20 mg pamiparib twice a day for the following 21 days (Day 3 to Day 23) until unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
- Phase 1: 40 mg Pamiparib: Participants received a single dose of 40 mg pamiparib orally on Day 1 followed by a one day treatment free period (Day 2), and 40 mg pamiparib twice a day for the following 21 days (Day 3 to Day 23) until unacceptable toxicities, disease progression, withdrawal of consent, investigator discretion, or delay of treatment due to unresolved toxicities for more than 21 days
Arm/Group | Phase 1: 20 mg Pamiparib | Phase 1: 40 mg Pamiparib | Phase 1: 60 mg Pamiparib | Phase 2: 60 mg Pamiparib in Platinum-sensitive Ovarian Cancer (PSOC) | Phase 2: 60 mg Pamiparib in Platinum-resistant Ovarian Cancer (PROC)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/7 | 37/90 | 18/23
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 2/7 | 36/90 | 15/23
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 7/7 | 90/90 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: 20 mg Pamiparib (N=4) | Phase 1: 40 mg Pamiparib (N=4) | Phase 1: 60 mg Pamiparib (N=7) | Phase 2: 60 mg Pamiparib in Platinum-sensitive Ovarian Cancer (PSOC) (N=90) | Phase 2: 60 mg Pamiparib in Platinum-resistant Ovarian Cancer (PROC) (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 16 (22) | 7 (11) — Adverse Events were coded based on MedDRA version 22.0 for Phase 1, and version 24.0 for Phase 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (2)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: 20 mg Pamiparib (N=4) | Phase 1: 40 mg Pamiparib (N=4) | Phase 1: 60 mg Pamiparib (N=7) | Phase 2: 60 mg Pamiparib in Platinum-sensitive Ovarian Cancer (PSOC) (N=90) | Phase 2: 60 mg Pamiparib in Platinum-resistant Ovarian Cancer (PROC) (N=23)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 2 (2) | 81 (204) | 21 (43)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erythropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 20 (71) | 3 (13)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (16) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (27) | 2 (15)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (13) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 5 (9) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 15 (25) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 10 (17) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (6) | 8 (11) | 1 (10)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (10) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 20 (40) | 6 (7)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Gastric dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (3) | 5 (11) | 61 (173) | 16 (34)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 2 (2) | 2 (4) | 46 (123) | 11 (47)
Asthenia (General disorders) | 3 (5) | 4 (5) | 5 (10) | 26 (36) | 6 (9)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (9) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 15 (30) | 2 (4)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 10 (11) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 17 (32) | 4 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (14) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 22 (38) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 24 (36) | 4 (6)
Bilirubin conjugated increased (Investigations) | 1 (5) | 1 (2) | 2 (4) | 5 (13) | 3 (6)
Bilirubin urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 6 (8) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (3) | 1 (1) | 0 (0) | 14 (46) | 4 (6)
Blood bilirubin unconjugated increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 4 (15) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 9 (10) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (11) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 2 (6) | 1 (3) | 2 (2) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (2) | 2 (2) | 16 (22) | 6 (6)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 5 (9) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 19 (49) | 5 (5)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (4) | 4 (5) | 57 (262) | 13 (57)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Neutrophil percentage increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 28 (78) | 10 (21)
Procalcitonin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Total bile acids increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Urine ketone body present (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 11 (13) | 4 (4)
White blood cell count decreased (Investigations) | 2 (2) | 3 (5) | 5 (8) | 55 (245) | 14 (41)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 3 (4) | 3 (9) | 30 (44) | 5 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2) | 3 (5) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (5) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 13 (25) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (10) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT03333915/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT03333915/SAP_001.pdf